CLINICAL TRIAL: NCT02667925
Title: Study of the Isotopic Distribution of Intraperitoneal Postoperative Locoregional Chemotherapy for Peritoneal Carcinomatosis of Ovarian Origin
Brief Title: Study of the Isotopic Distribution of Intraperitoneal Chemotherapy for Peritoneal Carcinomatosis of Ovarian Origin
Acronym: ISOTOVE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of the obsolescence of the study
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-004103-12
Record Dates: First submitted 2016-01-19; First posted 2016-01-29 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-09

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; intraperitoneal chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — nanocis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention arm (Experimental): Patients will receive an intraperitoneal chemotherapy (cisplatin) combined to a radiotracer (nanocis) in order to assess the intraperitoneal distribution of the chemotherapy
  Interventions: Drug: Intraperitoneal cisplatin with nanocis

INTERVENTIONS:
Drug: Intraperitoneal cisplatin with nanocis — Patients will receive an intraperitoneal chemotherapy combined to a radiotracer in order to assess the intraperitoneal distribution of the chemotherapy

SUMMARY:
The treatment of advanced ovarian cancer is based on the combination of chemotherapy based on platinum salt and surgery whose quality is the major prognostic factor.

A meta-analysis of retrospective series had shown that for every 10% increase in the complete cytoreduction rates were increased by 5.5% overall survival time (Markman et al, 2001). Currently, it is recognized that the best chance of survival conferred to patients whose initial surgical residue is zero (Harter et al, 2009).

However, even if macroscopically complete surgery and whatever the type of systemic chemotherapy, peritoneal recurrence remains high for more than 75%.

To reducing it of recurrence, a therapeutic approach is to administer chemotherapy intraperitoneally.

The intraperitoneal chemotherapy consists to administer the drug directly into the peritoneal cavity.

Alberts et al, 1996 and Armstrong et al, 2006 compared the efficacy in terms of survival of an intraperitoneal chemotherapy according to this method with a conventional systemic chemotherapy. Alberts reported a significant improvement in the median overall survival. Armstrong shows in addition a decreased risk of recurrence.

It must be remembered that:

* The establishment of an intra-abdominal catheter does not always ensure complete flow of drugs into the peritoneal cavity (major postoperative adhesions).
* There may be problems of catheters becoming blocked and requiring local treatment; these problems can cause abdominal pain whose care is difficult. Thus almost half of patients fail to get all six courses of intraperitoneal chemotherapy.

Thus, the investigators propose to estimate the flow of intraperitoneal chemotherapy with IP peritoneal scintigraphy, using a radiotracer (nanocis®). The investigators hypothesize that the movement of colloids in peritoneal cavity is similar to the circulation of chemotherapy within the peritoneal cavity (From Forni et al, 1993, Varia et al, 2003, Young et al, 2003, Dawson et al, 2011). The accumulation of radiotracer will be more correlated with abdominal pain sites described by the patient as well as peritoneal recurrence sites found during monitoring.

DETAILED DESCRIPTION:
Epithelial ovarian cancer is the fifth leading cause of female cancer and the leading cause of death among gynecological cancers (Alberts et al, 2002). The treatment of advanced ovarian cancer is based on the combination of chemotherapy based on platinum salt and surgery whose quality is the major prognostic factor.

A meta-analysis of retrospective series had shown that for every 10% increase in the complete cytoreduction rates were increased by 5.5% overall survival time (Markman et al, 2001). Currently, it is recognized that the best chance of survival conferred to patients whose initial surgical residue is zero (Harter et al, 2009).

However, even if macroscopically complete surgery and whatever the type of systemic chemotherapy, peritoneal recurrence remains high for more than 75%.

To reducing it of recurrence, a therapeutic approach is to administer chemotherapy intraperitoneally.

The intraperitoneal chemotherapy consists to administer the drug directly into the peritoneal cavity at a frequency that is related to systemic chemotherapy (every 3 weeks).

Alberts et al, 1996 and Armstrong et al, 2006 compared the efficacy in terms of survival of an intraperitoneal chemotherapy according to this method with a conventional systemic chemotherapy. Alberts reported a significant improvement in the median overall survival (49 vs 41 months). Armstrong shows in addition a decreased risk of recurrence.

It must be remembered that:

* The establishment of an intra-abdominal catheter does not always ensure complete flow of drugs into the peritoneal cavity (major postoperative adhesions).
* There may be problems of catheters becoming blocked and requiring local treatment; these problems can cause abdominal pain whose care is difficult. Thus almost half of patients fail to get all six courses of intraperitoneal chemotherapy.

Thus, the investigators propose to estimate the flow of intraperitoneal chemotherapy with IP peritoneal scintigraphy, using a radiotracer (nanocis®). The investigators hypothesize that the movement of colloids in peritoneal cavity is similar to the circulation of chemotherapy within the peritoneal cavity (From Forni et al, 1993, Varia et al, 2003, Young et al, 2003, Dawson et al, 2011). The accumulation of radiotracer will be more correlated with abdominal pain sites described by the patient as well as peritoneal recurrence sites found during monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Performance Status 0-2
* PNN> 1.5.109 / L (without added GCSF)
* Plaquettes> 100. 109 / L
* Bilirubine inferior or equal to 1.5 times the upper normal value (VNS)
* ASAT And ALT inferior or equal to 2.5 upper normal value (VNS)
* Alkaline Phosphatase inferior or equal to2.5 upper normal value (VNS)
* Clairance Creatinine> 60ml / min Normal -Ionogramme
* PTT <1.5 times the upper normal value (VNS) (heparin, or other accepted lovenox anticoagulants)
* PT / INR inferior or equal to 1.5 upper normal value (VNS) (or INR between 2 and 3, if the patient receives a stabilized dose of Warfarin)
* Patient operated first line without macroscopic residual for ovarian cancer or primary peritoneal or tubal stage IIIC or IV peritoneal pleural
* Minimum Required for surgery: hysterectomy, oophorectomy, pelvic lymphadenectomy and para-aortic omentectomy
* Patient requiring adjuvant chemotherapy
* Compulsory affiliation to a social security scheme.
* Obtaining informed consent in writing, signed and dated.

Exclusion Criteria:

* Patient with cognitive and psychiatric disorders.
* Patient deprived of liberty by a court or administrative.
* Patient having directions against the achievement of chemotherapy
* Concomitant treatment with a drug test, participation in another therapeutic clinical trial within 30 days
* Pregnant women
* Nursing women
* Patient with recognized hypersensitivity to cisplatin or platinum-containing products
* Patient with hypersensitivity recognized paclitaxel or any of the excipients
* Patient must be vaccinated against yellow fever
* Patient before taking phenytoin for prophylactic purposes
* Patient with hearing impairment
* Patient with hepatic impairment
* Patient with renal impairment Sensory or motor -Neuropathies> grade 1 (CTCAE)
* Hépatite Or severe infection requiring parenteral antibiotics
* Serious non-healing wound or ulcer, or bone fracture
* Fistule Abdominal or gastrointestinal perforation, or intra-abdominal abscess in the 28 days preceding the intraperitoneal chemotherapy Clinical -Symptômes, gastrointestinal obstruction or signs and / or which require a hydration and / or parenteral nutrition
* Patientes Has had or currently with inflammatory bowel disease
* Active bleeding or medical condition that carries a high risk of bleeding (eg, known coagulation disorders, coagulopathy, or tumor with large vessels)
* Cerebrovascular accident (CVA) or transient ischemic attack, or subarachnoid hemorrhage in the last 6 months
* Disease clinically significant cardiovascular, including:

  * uncontrolled hypertension, defined as systolic blood pressure> 150mmHg or diastolic> 90mmHg
  * myocardial infarction or unstable angina within the last 6 months
  * NYHA class II-IV congestive heart failure
  * serious cardiac arrhythmia requiring treatment: -an asymptomatic atrial fibrillation with controlled ventricular rate supraventricular tachycardia or controlled with medication and is authorized asymptomatic peripheral vascular disease o ≥ Grade 2 (CTCAE) (brief [less than 24 hours] ischemia episodes managed non-surgically and without permanent deficit)
* Antecedents of Hemorrhage or stroke (stroke), transient ischemic attack, or subarachnoid in the last 6 months Major Surgery within 28 days prior to inclusion

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Quantification by visual analysis the intensity of fixation of the solvent characterized in the intraperitoneal cavity | During the 6 cycles of chemotherapy, that is during 18 weeks
  The intensity of fixation will be defined as followed:
  0: no fixation
  1. fixation of low intensity
  2. fixation of high intensity

SECONDARY OUTCOMES:
Note adverse events assessed with CTCAE v4.0 | During the 6 cycles of chemotherapy, that is during 18 weeks
  The treatment-related adverse events will be assessed with CTCAE v4.0
Correlate pain intensity to fixation intensity in the peritoneal cavity | During the 6 cycles of chemotherapy, that is during 18 weeks
  Pain intensity will be measured with EVA scale
dosimetric study with peritoneal scintigraphy | During the 6 cycles of chemotherapy, that is during 18 weeks
  This study will be realised only for the first three patients included in the trial
Correlate site of relapse to localisation of labeled intraperitoneal solvent by nanocis in peritoneal cavity | During 5 years after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Pomel, MD, PhD, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harter P, Hilpert F, Mahner S, Kommoss S, Heitz F, Pfisterer J, du Bois A. Prognostic factors for complete debulking in first- and second-line ovarian cancer. Int J Gynecol Cancer. 2009 Dec;19 Suppl 2:S14-7. doi: 10.1111/IGC.0b013e3181bffb3f. PMID 19955907
- [Background] de Forni M, Boneu A, Otal P, Martel P, Shubinski R, Bugat R, Lucot H. Anatomic changes in the abdominal cavity during intraperitoneal chemotherapy: prospective study using scintigraphic peritoneography. Bull Cancer. 1993 Apr;80(4):345-50. PMID 8173187
- [Background] Varia MA, Stehman FB, Bundy BN, Benda JA, Clarke-Pearson DL, Alvarez RD, Long HJ; Gynecologic Oncology Group. Intraperitoneal radioactive phosphorus (32P) versus observation after negative second-look laparotomy for stage III ovarian carcinoma: a randomized trial of the Gynecologic Oncology Group. J Clin Oncol. 2003 Aug 1;21(15):2849-55. doi: 10.1200/JCO.2003.11.018. PMID 12885800
- [Background] Young RC, Brady MF, Nieberg RK, Long HJ, Mayer AR, Lentz SS, Hurteau J, Alberts DS. Adjuvant treatment for early ovarian cancer: a randomized phase III trial of intraperitoneal 32P or intravenous cyclophosphamide and cisplatin--a gynecologic oncology group study. J Clin Oncol. 2003 Dec 1;21(23):4350-5. doi: 10.1200/JCO.2003.02.154. PMID 14645424
- [Background] Dawson SJ, Hicks RJ, Johnston V, Allen D, Jobling T, Quinn M, Rischin D. Intraperitoneal distribution imaging in ovarian cancer patients. Intern Med J. 2011 Feb;41(2):167-71. doi: 10.1111/j.1445-5994.2009.02112.x. PMID 19849742
- [Background] Alberts DS, Liu PY, Hannigan EV, O'Toole R, Williams SD, Young JA, Franklin EW, Clarke-Pearson DL, Malviya VK, DuBeshter B. Intraperitoneal cisplatin plus intravenous cyclophosphamide versus intravenous cisplatin plus intravenous cyclophosphamide for stage III ovarian cancer. N Engl J Med. 1996 Dec 26;335(26):1950-5. doi: 10.1056/NEJM199612263352603. PMID 8960474
- [Background] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300